CLINICAL TRIAL: NCT07323940
Title: Correlation Between Multiscale Entropy Analysis of Electroencephalograms and Postoperative Delirium Incidence.
Brief Title: Correlation Between Perioperative EEG Variability and Postoperative Delirium Incidence.
Status: Recruiting | Type: Observational
Sponsor: Xin Chen (Other)
Collaborators: Second Affiliated Hospital of Hainan Medical College (Unknown)
Responsible Party: Sponsor-Investigator, Xin Chen, Associate Researcher,the Second Affiliated Hospital of Hainan Medical University, Hainan Medical College
Organization: Hainan Medical College (Other)
Other Study IDs: HUMU2H-EEGAMSE-CN-2025; No.823RC592 (Other Grant/Funding Number: Hainan Provincial Natural Science Foundation of China)
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Delirium - Postoperative
Keywords: Postoperative delirium; electroencephalogram; Multiscale Entropy
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly surgical patients undergoing general anaesthesia.
  Interventions: Device: Collect preoperative and intraoperative electroencephalogram data

INTERVENTIONS:
Device: Collect preoperative and intraoperative electroencephalogram data — Use Neuron-Spectrum-5-1 to collect preoperative and intraoperative electroencephalogram data.

SUMMARY:
This clinical study aims to investigate whether multiscale entropy analysis of electroencephalogram data can distinguish between ordinary elderly surgical patients and elderly patients with postoperative delirium.This study may help identify postoperative delirium in surgical patients at an early stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing general anaesthesia with single-lumen endotracheal tube placement;
2. Age ≥65 years, gender unrestricted, body mass index (BMI) 18-28 kg/m²;
3. Normal mouth opening and head/neck mobility;
4. Pre-anaesthesia American Society of Anaesthesiologists (ASA) physical status classification of I or II and Mallampati airway classification of I or II.

Exclusion Criteria:

1. Individuals with psychiatric disorders, literacy issues, or communication difficulties who are unable to cooperate with POD screening;
2. Patients with severe lesions in vital organs, such as the heart, lungs, brain, liver or kidneys.
3. Those undergoing cardiac or neurosurgical procedures during this admission;
4. A history of alcohol abuse or recent use of sedatives or opioids;
5. haemoglobin <100 g/L;
6. Participation in any clinical research studies within the past 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly surgical patients undergoing general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Within seven days after surgery(Day 0-7)
  Using the 3D-CAM scale to assess postoperative delirium in surgical patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology,the Second Affiliated Hospital of Hainan Medical University, Haikou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xu N, Li LX, Wang TL, Jiao LQ, Hua Y, Yao DX, Wu J, Ma YH, Tian T, Sun XL. Processed Multiparameter Electroencephalogram-Guided General Anesthesia Management Can Reduce Postoperative Delirium Following Carotid Endarterectomy: A Randomized Clinical Trial. Front Neurol. 2021 Jul 12;12:666814. doi: 10.3389/fneur.2021.666814. eCollection 2021. PMID 34322079
- [Result] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Result] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Aceto P, Audisio R, Cherubini A, Cunningham C, Dabrowski W, Forookhi A, Gitti N, Immonen K, Kehlet H, Koch S, Kotfis K, Latronico N, MacLullich AMJ, Mevorach L, Mueller A, Neuner B, Piva S, Radtke F, Blaser AR, Renzi S, Romagnoli S, Schubert M, Slooter AJC, Tommasino C, Vasiljewa L, Weiss B, Yuerek F, Spies CD. Update of the European Society of Anaesthesiology and Intensive Care Medicine evidence-based and consensus-based guideline on postoperative delirium in adult patients. Eur J Anaesthesiol. 2024 Feb 1;41(2):81-108. doi: 10.1097/EJA.0000000000001876. Epub 2023 Aug 30. PMID 37599617